CLINICAL TRIAL: NCT07165717
Title: A Real World Study of Respiratory Critical Disease.
Status: Recruiting | Type: Observational
Sponsor: Ming Zhong (Other)
Responsible Party: Sponsor-Investigator, Ming Zhong, PI, Shanghai Zhongshan Hospital
Organization: Shanghai Zhongshan Hospital (Other)
Other Study IDs: B2023-016
Record Dates: First submitted 2025-06-13; First posted 2025-09-10 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: ARDS (Acute Respiratory Distress Syndrome); Real World Study
MeSH Terms: conditions — Acute Lung Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No Intervention: Observational Cohort — Obsercational study

SUMMARY:
Acute Respiratory Distress Syndrome (ARDS) is a form of acute diffuse lung injury caused by various etiologies, which rapidly progresses to acute respiratory failure. It is characterized by a sudden onset and severe clinical course. Globally, ARDS affects approximately 3 million individuals each year, accounting for about 10% of admissions to intensive care units (ICUs). Due to the lack of specific pharmacological therapies, mechanical ventilation remains the mainstay of treatment. Therefore, identifying and analyzing prognostic factors for ARDS patients is of great significance for improving patient outcomes and reducing the incidence of poor prognosis.

ELIGIBILITY:
Inclusion Criteria:

* Patients with underlying diseases associated with high risk of ARDS, including but not limited to: sepsis, pneumonia, multiple trauma, pulmonary contusion, inhalation injury, massive blood transfusion, other high-risk conditions, or other factors causing excessive respiratory drive.
* Patients meeting the inclusion criteria for a high-risk ARDS population.
* Patients (or legal representatives) who have provided a signed and dated informed consent form.

Exclusion Criteria:

* Age under 18 years.
* HIV infection.
* Known immunodeficiency disorders (e.g., leukemia, common variable immunodeficiency, etc.).
* History of solid organ or bone marrow transplantation.
* Receiving treatment with G-CSF or GM-CSF.
* Patients with a decision to withdraw from active treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients identified as high risk for ARDS after ICU admission.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2019-03-01 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Mortality | Day 28 after ARDS diagnosis
  Clinical observation
Mortality | Day 60 after ARDS diagnosis
  Clinical observation

SECONDARY OUTCOMES:
Chest CT Scan | Monitored daily
  Chest CT imaging
Complete Blood Count | Monitored daily
  Blood sampling and laboratory testing
Serial Arterial Blood Gas Monitoring | Monitored daily after enrollment
  Arterial blood gas collection
Fluid Input and Output Balance | Whenever fluid input or output occurs
  Clinical nursing records
Mechanical Ventilation Monitoring | Every second after intubation
  Automatically recorded by ventilator

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University, Zhong Shan Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes